CLINICAL TRIAL: NCT02426190
Title: Knee Arthroplasty Rehabilitation Outcomes Study
Acronym: KAROS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MedStar National Rehabilitation Network (Other)
Responsible Party: Principal Investigator, Jean Hsieh, PhD, Senior Research Associate, MedStar National Rehabilitation Network
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012-347
Record Dates: First submitted 2015-04-08; First posted 2015-04-24 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Total Knee Arthroplasty; Rehabilitation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 (Active Comparator): Patients in Arm 1 receive standard of care rehabilitation protocol using a recumbent or Nu-step bike during warm-up, followed by individualized therapeutic exercise, and cool-down protocols. The warm-up phase in the study refers to therapeutic exercise. The therapeutic exercise aims to condition and prepare patients for subsequent functional or therapeutic activities. The active comparator (Arm 1) is to ask participants to use modalities, such as a recumbent bike or a Nu-step bike during the warm-up phase of an outpatient physical therapy following a single total knee replacement.
  Interventions: Other: Recumbent or Nu-step bike
- Arm 2 (Experimental): Patients in Arm 2 will use an anti-gravity treadmill (AlterG) during warm-up, followed by individualized therapeutic exercise and cool-down protocols.
  Interventions: Other: Anti-gravity treadmill
- Arm 3 (Experimental): Patients in Arm 3 will use a recumbent or Nu-step bike along with the PENS neuromuscular stimulation modality during warm-up, followed by individualized therapeutic exercise and cool-down protocols.
  Interventions: Other: PENS - neuro-muscular stimulation
- Arm 4 (Experimental): Patients in Arm 4 will use both an anti-gravity treadmill (AlterG) and the PENS neuromuscular stimulation modality during warm-up, followed by individualized therapeutic exercise and cool-down protocols.
  Interventions: Other: Anti-gravity treadmill & PENS - neuro-muscular stimulation

INTERVENTIONS:
Other: Anti-gravity treadmill — The intervention is to ask study participants to ambulate using an anti-gravity treadmill that integrates patented, NASA Differential Air Pressure (DAP) technology -- a precise air calibration system -- to uniformly reduce gravitational load and body weight during the warm-up phase of an outpatient physical therapy following a single total knee replacement.
  Arms: Arm 2
Other: PENS - neuro-muscular stimulation — The intervention is to ask study participants to warm up using Patterned Electrical Neuromuscular Stimulation (PENS) - that closely replicates the body's normal muscle and nerve firing patterns -- on his/her surgical leg in conjunction with a recumbent bike or a Nu-step bike during the warm-up phase of an outpatient physical therapy following a single total knee replacement.
  Arms: Arm 3
Other: Anti-gravity treadmill & PENS - neuro-muscular stimulation — The intervention is to ask study participants to ambulate using an anti-gravity treadmill in conjunction with use of Patterned Electrical Neuromuscular Stimulation (PENS) during the warm-up phase of an outpatient physical therapy following a single total knee replacement.
  Arms: Arm 4
Other: Recumbent or Nu-step bike — This is the active comparator of the trial that participants are asked to use either a recumbent or Nu-step bike normally seen in an outpatient physical therapy clinic to warm-up during a physical therapy session following a single total knee replacement.
  Arms: Arm 1

SUMMARY:
The objective of the KAROS study is to compare rehabilitation outcomes between 3 proposed protocols and a current standard of care protocol for the purpose of identifying better practice for outpatient rehabilitation among patients with single total knee replacement. The 3 advanced protocols involve use of an anti-gravity treadmill and/or the patterned electrical neuromuscular stimulation (PENS). Both medical modalities have been cleared by the FDA to be used in medical rehabilitation, including total knee replacement.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo an elective single total knee arthroplasty and initiate their outpatient rehabilitation therapy within 3 weeks after surgery.
* Patients who are 40 years old or older.
* Patients who weight less than 320 lb to accommodate the weight limit to use the anti-gravity treadmill.

Exclusion Criteria:

* Patients who had any lower extremity joint replacement less than 1 year prior the current total knee replacement.
* Patients who are pregnant or may be pregnant.
* Patients who have a medical history of neurologic disorders.
* Patients who have received more than 2 weeks of other formats of rehabilitation prior their outpatient rehabilitation program.
* Patients who received any cancer treatment in the past year prior the current surgery.
* Patients who have uncontrolled cardiovascular hypertension.
* Patients who have cardiac demand pacemakers and/or implanted defibrillators.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 386 (Actual)
Dates: Start 2014-10; Primary Completion 2017-12 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
AM-PAC (Activity Measure for Post Acute Care) Basic Mobility score: Baseline | Baseline
  The primary outcome measure is the AM-PAC Basic Mobility score. AM-PAC is a patient-reported instrument to measure functional level in 3 domains: basic mobility, daily activity, and applied cognition. For the purpose of the study, only the basic mobility domain was measured. Using item-response theory, the AM-PAC program selects the most representative questions from its extensive item bank to ask when measuring a patient's functional level. This study used the AM-PAC basic mobility paper short form designed for outpatient settings. The short-form consists of 18 questions and produces a raw score (18 to 72) transformed into a score ranging from 29.41 to 80.30 based on item-degree of difficulty. Higher transformed scores denote higher functional mobility: 34 - 51.9 = limited indoor mobility; 52 - 65.9 = enhanced indoor mobility; 66 and above = outdoor mobility.
AM-PAC (Activity Measure for Post Acute Care) Basic Mobility score: Discharge from outpatient rehabilitation | Discharge from outpatient rehabilitation (on average 2 months from baseline)
  The primary outcome measure is the AM-PAC Basic Mobility score upon discharge from outpatient therapy. AM-PAC is a patient-reported instrument to measure functional level in 3 domains: basic mobility, daily activity, and applied cognition. For the purpose of the study, only the basic mobility domain was measured. Using item-response theory, the AM-PAC program selects the most representative questions from its extensive item bank to ask when measuring a patient's functional level. This study used the AM-PAC basic mobility paper short form designed for outpatient settings. The short-form consists of 18 questions and produces a raw score (18 to 72) transformed into a score ranging from 29.41 to 80.30 based on item-degree of difficulty. Higher transformed scores denote higher functional mobility: 34 - 51.9 = limited indoor mobility; 52 - 65.9 = enhanced indoor mobility; 66 and above = outdoor mobility.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Vita, DPT, Principal Investigator — MedStar National Rehabilitation Network
Locations (1):
- MedStar National Rehabilitation Network, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Hsieh CJ, DeJong G, Vita M, Zeymo A, Desale S. Effect of Outpatient Rehabilitation on Functional Mobility After Single Total Knee Arthroplasty: A Randomized Clinical Trial. JAMA Netw Open. 2020 Sep 1;3(9):e2016571. doi: 10.1001/jamanetworkopen.2020.16571. PMID 32940679
- [Derived] DeJong G, Hsieh CJ, Vita MT, Zeymo A, Boucher HR, Thakkar SC. Innovative Devices Did Not Provide Superior Total Knee Arthroplasty Outcomes in Post-Operative Rehabilitation: Results From a Four-Arm Randomized Clinical Trial. J Arthroplasty. 2020 Aug;35(8):2054-2065. doi: 10.1016/j.arth.2020.03.048. Epub 2020 Apr 2. PMID 32360105